CLINICAL TRIAL: NCT03082612
Title: Faith-Based African American Cancer Survivorship Storytelling: A Culturally Relevant Intervention to Alleviate Psychological Stress
Brief Title: Faith-Based African American Cancer Survivorship Storytelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jill Hamilton, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00093110; 5R03MD013509-02 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-03-17 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Behavioral research; Social research; Spirituality; Late stage cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- African American cancer patients (Experimental): Patients will be required to participate in intervention activities and 5 data collection interviews. Interviews to complete both open-ended interviews and quantitative measures will take approximately 45 minutes. The actual administration of the intervention (viewing of video recordings) will take approximately 30 minutes with all sessions to occur over a 3 week period.
  Interventions: Behavioral: Faith-Based African American Cancer Survivorship Storytelling Intervention
- Family caregivers (Experimental): Family caregivers will be required to participate in intervention activities and 5 data collection interviews. Interviews to complete both open-ended interviews and quantitative measures will take approximately 45 minutes. The actual administration of the intervention (viewing of video recordings) will take approximately 30 minutes with all sessions to occur over a 3 week period.
  Interventions: Behavioral: Faith-Based African American Cancer Survivorship Storytelling Intervention

INTERVENTIONS:
Behavioral: Faith-Based African American Cancer Survivorship Storytelling Intervention — The intervention will consist of participants viewing a selection of video recorded vignettes during 3 weekly sessions. There will be 5 vignettes included in each session with each vignette edited to a real time of 3-4 minutes (each session is 30 minutes). Since the intervention is designed to be self-administered, there will be a video recorded introduction and instructions for use narrated by the PI. The vignettes are of actual African American cancer survivors narrating stories of ways in which hymns can be used to overcome their anxieties and depressed moods through the use of a hymn. The hymns included represent exemplars from the 5 themes prevalent in the PI's previous research
  Other Names: Hymns Intervention

SUMMARY:
The purpose of this research study is to evaluate the feasibility and acceptability of an intervention (viewing of video recordings) designed to reduce psychological distress among African Americans during treatment for cancer. This knowledge will inform a larger test of an intervention.

DETAILED DESCRIPTION:
This study addresses a need to integrate spirituality with cancer care as requested among African Americans. In the PI's research with African Americans, a dominant mental health promoting strategy used in response to a cancer diagnosis is the use of religious stories and songs. African Americans have a strong cultural history of relying on religious stories and songs to overcome oppression and mental suffering encountered in their lived experience. If successful, the findings from this preliminary study will contribute to the evidence that spirituality is important to cancer care and to achieving optimal patient outcomes among this medically underserved population. More importantly, the infusion of spirituality in cancer care has to potential to reduce the high levels of psychological distress experienced among African Americans and FCG's; to enable them to become more engaged in their cancer care and in supportive family relationships; and, ultimately to improve the overall quality of life for African American cancer patients and FCGs. The actual administration of the intervention (viewing of video recordings) will take approximately 30 minutes with all sessions to occur over a 3 week period. The intervention will consist of participants viewing a selection of video recorded vignettes during 3 weekly sessions. The vignettes are of actual African American cancer survivors narrating stories of ways in which hymns can be used to overcome their anxieties and depressed moods through the use of a hymn.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Age 30-89 years
* Newly diagnosed with any stage cancer
* Treatment plans to include weekly outpatient chemotherapy
* Previously screened and with greater than 0 level of psychological distress
* Willingness to participate in all study activities including data collection
* Willing to identify a family caregiver (FCG) (immediate or extended family member) to also participate

Exclusion Criteria for Patients:

* Have completed surgery with no plans for chemotherapy
* Find conversations around religion or spirituality emotionally upsetting
* Have completed more than half of prescribed chemotherapy treatments
* In hospice care
* Not able to provide informed consent

Inclusion Criteria for Family Caregiver:

* Immediate or extended family member of the patient
* 18 years of age or older
* Able to provide informed consent
* Willing to participate in study activities, including data collection

Exclusion Criteria for Family Caregiver:

* Find conversations around religion or spirituality emotionally upsetting

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill B Hamilton, PhD, RN, Principal Investigator — Emory University
Locations (1):
- Grady Cancer Center for Excellence, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total enrollment number represents the number of individual participants including African American Cancer patients and Family caregivers.
Period: Overall Study
Arm/Group | African American Cancer Patients | Family Caregivers
Started | 17 | 5
Completed | 15 | 5
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African American Cancer Patients | Family Caregivers | Total
Number analyzed (Participants) | 17 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (15.8) | 46.4 (14.3) | 54.27 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 3 | 20
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 5 | 22
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety and Depression Scale (HADS) Score
Description: Psychological distress for patients and family caregivers (FCGs) will be measured with the Hospital Anxiety and Depression Scale (HADS).
  Scoring for the Anxiety and Depression scale of the HADS is (0-21); Normal (0-7); Borderline Abnormal Case (8-10); and Abnormal Case (11-21). Higher score correlates with worse outcome.
Time Frame: Baseline, Week 3 post-intervention
Population: Number of participants analyzed include participants that completed the Hospital Anxiety and Depression Scale (HADS) in the study sessions for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- African American Cancer Patients and Family Caregivers: Patients will be required to participate in intervention activities and 5 data collection interviews. Interviews to complete both open-ended interviews and quantitative measures will take approximately 45 minutes. The actual administration of the intervention (viewing of video recordings) will take approximately 30 minutes with all sessions to occur over a 3 week period.
  Faith-Based African American Cancer Survivorship Storytelling Intervention: The intervention will consist of participants viewing a selection of video recorded vignettes during 3 weekly sessions. There will be 5 vignettes included in each session with each vignette edited to a real time of 3-4 minutes (each session is 30 minutes). Since the intervention is designed to be self-administered, there will be a video recorded introduction and instructions for use narrated by the PI. The vignettes are of actual African American cancer survivors narrating stories of ways in which hymns can be used to overcome their anxieties and depressed moods through the use of a hymn. The hymns included represent exemplars from the 5 themes prevalent in the PI's previous research
Arm/Group | African American Cancer Patients and Family Caregivers | Family Caregivers
Number analyzed (Participants) | 15 | 5
score on a scale
  Baseline | 3.86 (2.53) | 0.60 (0.54)
  Week 3 post-intervention | 3.40 (3.22) | 1.20 (1.30)

2. Secondary Outcome: Supportive Family Relationships (Mutuality) Scale Score
Description: Mutuality is measured with the scale "You, Your Family and Friends" that measures the degree of positive relationships among participants and their family and friends. This scale measures the degree to which the caregiver-care receiver relationship was characterized by love, shared values, shared pleasurable activities, and reciprocity. The adapted scale has 12-items with a 5-point response format. A mean of responses with a range of 0 to 5 will be reported. Higher scores are indicative of better outcomes, indicating engagement in positive supportive relationships with family and friends.
Time Frame: Baseline, Week 3 post-intervention
Population: Number of participants analyzed include participants that completed the Supportive Family Relationships (Mutuality) Scale in the study sessions for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Cancer Patients and Family Caregivers | Family Caregivers
Number analyzed (Participants) | 15 | 5
score on a scale
  Baseline | 3.53 (0.46) | 3.34 (0.82)
  Week 3 post-intervention: number analyzed (Participants) | 14 | 5
  Week 3 post-intervention | 3.48 (0.41) | 3.50 (0.53)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 weeks.
Arm/Group | African American Cancer Patients | Family Caregivers
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/5
Other Adverse Events (participants affected / at risk) | 0/17 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03082612/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03082612/ICF_000.pdf